CLINICAL TRIAL: NCT00944541
Title: Pilot Study Evaluating Maraviroc (Celsentri®)Intensification Benefit in HIV Infected Patients Presenting Insufficient Immune Restoration Despite Controlled Viral Load With Antiretroviral Treatment. ANRS 145 MARIMUNO
Brief Title: Evaluation of Maraviroc Intensification in HIV Infected Patients With Insufficient Immune Restoration
Acronym: 145 MARIMUNO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2009-011171-76; ANRS 145 MARIMUNO
Record Dates: First submitted 2009-07-22; First posted 2009-07-23 (Estimated); Last update posted 2011-12-22 (Estimated); Status verified 2011-12

CONDITIONS: HIV Infection; HIV Infections
Keywords: maraviroc; immune restoration; treatment intensification
MeSH Terms: conditions — HIV Infections | interventions — Maraviroc

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: maraviroc — maraviroc 150 mg or 300 mg or 600 mg twice a day for 24 weeks
  Other Names: Celsentri

SUMMARY:
This pilot study aims to evaluate Maraviroc intensification strategy during 24 weeks in HIV infected patients under efficient (CV< 50 cp/mL), controlled antiretroviral therapy (≥ 6 months) and uncompleted immune restoration (CD4<350 cells/mL and CD4 earning <100 cells/mL during last 24 months).

The study will include 60 patients whose follow up is carried out for 48 weeks. recruitment period will be maintained for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection
* maraviroc-naives patients
* CD4 less than 350 cells/mm3
* viral load less than 50 cp/mL and CD4 earning less than 100 cells/mm3 during last 24 months

Exclusion Criteria:

* HIV-2 infection
* X4 tropism at inclusion
* pregnancy and breast feeding
* interferon, immunomodulatory drugs treatment or anti-HIV vaccines and chemotherapy
* hypersensibility of peanut or soya

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-09; Primary Completion 2010-08 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of maraviroc intensification during 24 weeks in HIV infected patients with insufficient immune restoration despite controlled viral load | immunologic benefit at week 24

SECONDARY OUTCOMES:
Maraviroc efficacy at W24 (virological and immunological efficacy); Durability of maraviroc efficacy between W24 & W36; Cmin of maraviroc and other molecules at W4,12,24; Evaluation of the safety of maraviroc between W0 and W36. | immuno-virologic evolution between week 0 and week 36

CONTACTS AND LOCATIONS:
Overall Officials: Lise CUZIN, MD, Principal Investigator — CHU Purpan - Toulouse (France)
Locations (1):
- French National Agency for Research on AIDS and Viral Hepatits, Paris, France